CLINICAL TRIAL: NCT02191488
Title: Quantification of ALA-induced PpIX Fluorescence During Brain Tumor Resection
Brief Title: ALA-induced PpIX Fluorescence During Brain Tumor Resection
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David W. Roberts (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, David W. Roberts, Professor of Surgery (Neurosurgery), Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMS 13066; R01NS052274-01A2 (NIH)
Record Dates: First submitted 2014-07-09; First posted 2014-07-16 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Brain Tumors
Keywords: Fluorescence; Brain Tumors; Brain Metastases; Malignant Glioma; Brain Lesions
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: 5-aminolevulinic acid (Experimental): 20mg/kg 3 hours prior to surgery
  Interventions: Drug: 5-aminolevulinic acid

INTERVENTIONS:
Drug: 5-aminolevulinic acid
  Other Names: 5-ALA

SUMMARY:
Removing a tumor from a patients brain is hard to do because, very often, brain tumors do not have boundaries that are easy for the patients surgeon to find. In many cases, the surgeon can't tell exactly where the tumor begins or ends. The surgeon usually can remove most of the patient's tumor by looking at the MRI images that were taken of the patient's brain before surgery. However, the surgeon does not have any good way to tell if the entire tumor has been removed or not. Removing the entire tumor is very important because leaving tumor behind may allow it to grow back which could decrease the chances of survival.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative diagnosis of either presumed first-time low or high grade glioma, or recurrent glioma, or metastasis, or meningioma
* Tumor judged to be suitable for open cranial resection based on preoperative imaging studies.
* Patient or LAR able to provide written informed consent.
* No serious associated psychiatric illnesses.
* Age > 21 years old.

Exclusion Criteria:

* Pregnant women or women who are breast feeding
* History of cutaneous photosensitivity, porphyria, hypersensitivity to porphyrins, photodermatosis, exfoliative dermatitis.
* History of liver disease within the last 12 months.
* Elevated liver function levels greater than 2.5 times the normal limit from laboratory tests conducted within 30 days prior to surgery.
* Inability to comply with the photosensitivity precautions associated with the study.
* Plasma creatinine in excess of 180umol/L within 30 days prior to surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of intraoperative measurements of PpIX concentration to coregistered histopathology | Up to five years from the first surgery date
  To estimate the probability of tumor distribution for a given PpIX concentration by comparing intraoperative measurements with coregistered histopathology obtained from biopsy sampling during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: David W. Roberts, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Roberts DW, Olson JD, Evans LT, Kolste KK, Kanick SC, Fan X, Bravo JJ, Wilson BC, Leblond F, Marois M, Paulsen KD. Red-light excitation of protoporphyrin IX fluorescence for subsurface tumor detection. J Neurosurg. 2018 Jun;128(6):1690-1697. doi: 10.3171/2017.1.JNS162061. Epub 2017 Aug 4. PMID 28777025